CLINICAL TRIAL: NCT03398382
Title: Effect of Oral Magnesium Supplementation on Anesthesia and Postoperative Analgesia After Surgical Removal of the Lower Third Molars.
Brief Title: Effect of Oral Magnesium on Anesthesia and Postoperative Analgesia After Surgical Removal of the Lower Third Molars.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daniel Jerković (Other)
Responsible Party: Sponsor-Investigator, Daniel Jerković, Principal investigator, University of Zagreb
Organization: University of Zagreb (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 05-PA-15-3/2017
Record Dates: First submitted 2018-01-07; First posted 2018-01-12 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-01

CONDITIONS: Postoperative Pain; Third Molar; Postoperative Complications
Keywords: Magnesium citrate; Trismus after surgical removal of the lower third molars; Local anesthesia; Analgesia after surgical removal of the lower third molars; Swelling after surgical removal of the lower third molars; Surgical removal of the lower third molars; Oral surgical procedures; Placebo effect
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The study will be a double-blind, randomized, split mouth, placebo controlled trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The selection of anaesthesia combination with oral placebo or magnesium for each side will be determined by random selection, which will not be known to either the patient or the examiner until the trial is completed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Magnesium citrate tablet group (Placebo Comparator): In this group patients will take magnesium citrate tablets 3 days postoperatively, so 400 mg magnesium citrate tbl (Solgar) /per day will be taken at the same time that will correspond to the time the first tablets were taken, 2 hours preoperatively.
  Interventions: Dietary Supplement: Magnesium tablet group
- Placebo tablet group (Placebo Comparator): In this group patients will take placebo tablets 3 days postoperatively, so 400 mg /per day placebo tbl will be taken at the same time that will correspond to the time the first tablets were taken, 2 hours preoperatively.
  Placebo tablets will be identical to the right drug (Magnesium citrate tbl.Solgar)
  Interventions: Dietary Supplement: Placebo tablets group
- Magnesium citrate lozenge group (Placebo Comparator): In this group patients will take 100 mg. magnesium citrate lozenge (Diasporal) 30 min. before the procedure and continue to take up to 4 lozenges per day over the next 3 days in the same time intervals as it was on the day of surgery.
  Interventions: Dietary Supplement: Magnesium lozenge group
- Placebo lozenge group (Placebo Comparator): In this group patients will take 100 mg. placebo lozenge 30 min. before the procedure and continue to take up to 4 pastilles per day over the next 3 days in the same time intervals as it was on the day of surgery.
  Placebo lozenges will be identical to the right drug (Magnesium citrate tbl.(Diasporal)
  Interventions: Dietary Supplement: Placebo lozenges group

INTERVENTIONS:
Dietary Supplement: Magnesium tablet group — Before the anaesthesia, all principles of surgical sterility and asepsis with oral cavity flushing for 1 min. ( 15 ml. 0.12% CHX.) will be performed. Operative side will be anaesthetized with the same anaesthetic 3M ESPE, Ubistesin-artikain. The surgeon, assistant, surgical approach, surgery technique and instruments will be the same in all subjects. For one side which will be randomly selected, the patient will receive magnesium citrate tablets. The same analgesics will also be prescribed: Ibuprofen tbl 400 mg which will be taken as needed, and magnesium citrate tablets. 200 mg. After the surgery, all patients will be given the same written and oral instructions for postoperative care.
  Arms: Magnesium citrate tablet group
Dietary Supplement: Placebo tablets group — Before the anaesthesia, all principles of surgical sterility and asepsis with oral cavity flushing for 1 min. ( 15 ml. 0.12% CHX.) will be performed. Operative side will be anaesthetized with the same anaesthetic 3M ESPE, Ubistesin-articain. The surgeon, assistant, surgical approach, surgery technique and instruments will be the same in all subjects. For one side which will be randomly selected , the patient will receive placebo tablets which will be identical to the right drug. The same analgesics will also be prescribed: Ibuprofen tbl 400 mg which will be taken as needed, and placebo tablets. 200 mg. After the surgery, all patients will be given the same written and oral instructions for postoperative care.
  Arms: Placebo tablet group
Dietary Supplement: Magnesium lozenge group — Before the anaesthesia, all principles of surgical sterility and asepsis with oral cavity flushing for 1 min. ( 15 ml. 0.12% CHX..) will be performed. Operative side will be anaesthetized with the same anaesthetic 3M ESPE, Ubistesin-articain. The surgeon, assistant, surgical approach, surgery technique and instruments will be the same in all subjects. For one side which will be randomly selected patient will receive magnesium citrate lozenge.The same analgesics will also be prescribed: Ibuprofen tbl 400 mg which will be taken as needed, and magnesium citrate lozenges. 100 mg. After the surgery, all patients will be given the same written and oral instructions for postoperative care.
  Arms: Magnesium citrate lozenge group
Dietary Supplement: Placebo lozenges group — Before the anaesthesia, all principles of surgical sterility and asepsis with oral cavity flushing for 1 min. ( 15 ml. 0.12% CHX.) will be performed. Operative side will be anaesthetized with the same anaesthetic 3M ESPE, Ubistesin-articain. The surgeon, assistant, surgical approach, surgery technique and instruments will be the same in all subjects. For one side which will be randomly selected patient will receive placebo lozenges which will be identical to the right drug. The same analgesics will also be prescribed: Ibuprofen tbl 400 mg which will be taken as needed, and placebo lozenges 100 mg. After the surgery, all patients will be given the same written and oral instructions for postoperative care.
  Arms: Placebo lozenge group

SUMMARY:
The operation of the lower third molars is one of the most common oral surgery procedures in the world. The surgery is mostly done in local anesthesia which makes the surgery as pleasant as possible for the patient. In addition to anesthesia control, it is also extremely important to insure postoperative pain control since that is the nuisance that patients are most likely to complain about after oral surgery. It has been noticed that magnesium added to local anesthetics can improve and prolong its effect, but also reduce postoperative pain and accelerate recovery. It can also be used as an auxiliary to control pain and inflammation, which is why we will use it in this study, because we have not been able to find magnesium data in the literature for the removal of the lower third molars.

Studies that have already been conducted with oral magnesium are for the purpose of preventing asthma, migraine, for reducing mood swings in PMS, reducing pain after endotracheal intubation, and many others.

Removal by using operative procedure is the only way to remove lower third molars.

The main objective of the study is to demonstrate the influence of the orally received magnesium citrate (before and after surgical removal of the lower third molar) on the quality and duration of the anesthetic block and also its effect on postoperative pain control. Other specific objectives are to investigate the effect of pre/postoperatively received magnesium on:

1. swelling stage after surgery.
2. time occurrence and duration of anesthesia.
3. trismus stage after the operative procedure.
4. the total amount of analgetics taken after surgery Benefits for the respondents will be in the assumption that the anesthetic block of the mandibular nerve will last longer with better quality, thus making the surgical procedure more pleasant and that the overall postoperative pain will be lessened and recovery faster in the magnesium citrate group. We also assume that in the magnesium citrate group trismus will be less pronounced and that swelling in postoperative days will be smaller.

DETAILED DESCRIPTION:
Study design and sample description of this study was performed at the Department of Oral Surgery of Clinical Hospital Dubrava, Zagreb, Croatia.

Respondents are the patients who need to do the operation of both lower third molars and due to this they are in the Clinical Hospital Dubrava. All participants will sign informed consent for participation in the research. Their participation will be voluntary.

The study is approved by Ethics Committee of the School of Dental Medicine, Zagreb, Croatia (03.2017). The identity of the subjects will be protected in all phases of the study.

Respondents in this research will be exposed to the following risks:

Risks related to the procedure: pain, swelling, trismus, inflammation, paresthesia of the mandibular nerve branches (alveolar, lingualis), bleeding.

Drug related risks: allergic reactions, gastrointestinal symptoms (diarrhea). The study will be a double-blind, randomized, split mouth, placebo controlled trial.

It will be carried out with two different oral forms of magnesium citrate:

1. in tablet form,
2. in the form of a lozenge. Each of these forms will have a same group

1- tablet group, 2-lozenge group. Both of these groups will have a control placebo group. Before the anaesthesia, all principles of surgical sterility and asepsis with oral cavity flushing for 1 min. ( 15 ml. 0.12% CHX.-Chlorhexidine) will be performed Both sides (over a period of 14 days) will be anaesthetized with the same anaesthetic 3M ESPE, Ubistesin-articain (1ml injection suspension containing 40mg of articainchloridum and 0.005mg adrenalin in a form of adrenalinchloridium).

For one side, which will be randomly selected, the patient will receive magnesium citrate tablets (Solgar tablets) / lozenges (Diasporal lozenges), and for other placebo tablets / lozenges, which will be identical to the right drug, so the same examinee will be a test and control group. The surgeon, assistant, surgical approach, surgery technique and instruments will be the same in all subjects regardless of magnesium citrate or placebo group of the same.

The selection of anaesthesia combination with oral placebo or magnesium for each side will be determined by random selection, which will not be known to either the patient or the examiner until the test is completed. After the surgery, all patients will be given the same written and oral instructions for postoperative care.

The same analgesics will also be prescribed: Ibuprofen tbl 400 mg which will be taken as needed, and magnesium citrate tbl. 200 mg / magnesium citrate lozenges 100 mg or placebo depending on randomized selection.

Magnesium citrate tablets /placebo tablets patients will take 3 days postoperatively so that 400 mg /per day magnesium citrate tbl (Solgar) / placebo will be taken at the same time that will correspond to the time taken for the first tablets, 2 hours preoperatively.

In the group that will use lozenges the patients will take them 30 min. before the procedure a 100 mg. magnesium citrate lozenge (Diasporal) / placebo lozenge and continue to take up to 4 pastilles per day over the next 3 days in the same time intervals as it was on the day of surgery.

Therapeutic drug doses will be used far below the doses used in the previous studies where the magnesium citrate tablets were used.

During the use of magnesium citrate / placebo (3 days after surgery) the patient will fill out a prepared written questionnaire that will be discussed thoroughly before the first operation.

Postoperative follow-up will be done by the single experienced therapist and by the patient (see Outcome Measures).

The following symptoms which will be assessed are: pain, swelling, maximum inter-incisal opening of mouth, total amount of analgesics taken after surgery, time occurrence and duration of anesthesia and personal experience of pain after surgery (see Outcome Measures). These symptoms will be evaluated on the day of operation and 3 days after surgery.

The planned sample size is at least 40 molars in each group, that is 80 operations in a total of 40 patients using tablets, and equal to the group using lozenges.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 30 years of age (both gender)
* ASA1 (a normal healthy patient)
* Parant 3 (extraction requiring osteotomy and coronal section)
* non-dietary intake
* non-therapeutic
* no magnesium and anaesthetic allergies
* no analgesics taken in the last 24 hours
* without inflammations in the area
* lower third molars which have an identical position in bone

Exclusion Criteria:

* pregnant women
* breastfeeding women
* people on specific nutrition
* people with natural or acquired pathological conditions
* persons known for drug abuse analgesics or any kind of drugs
* patients who will use antibiotics or another drugs during postoperative recovery

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain | First 3 days after surgery
  Patients will evaluate their postoperative pain with grades from 0-10 according to visual analogue scale (VAS) where the end points were marked as "no pain" (0) and "unbearable pain"(10).
Duration of local anesthesia | During the first day of operation
  We will measure the time from the onset of anesthesia activity and the patient will write down when the activity of anesthesia has finished.

SECONDARY OUTCOMES:
Swelling stage after surgery | First 3 days after surgery
  The patient will get a prepared written questionnaire that will be discussed thoroughly before the first operation.
  For the swelling we will use a subjective evaluation scale with 4 parameters: none (no swelling), light (intraoral, localized to the treated area), moderate (extraoral swelling localized to the treated area), and severe (extraoral swelling extending beyond the treated area). Swelling will be determined during the first, second and third postoperative day by the patient.
Trismus stage after the operative procedure. | First 3 days after surgery
  The maximum inter-incisal opening of the mouth was calculated from the mesioincisal angle of the ipsilateral mandibular central incisor to the mesioincisal angle of the ipsilateral mandibular central incisor using the : TheraBite measure

OTHER OUTCOMES:
Patient's personal experience of the operation | On the day of operation
  Using VAS scale, we will determine the patient's personal experience of the operation

CONTACTS AND LOCATIONS:
Locations (2):
- Croatia (2):
  - Clinical Department of Oral Surgery, University Hospital "Dubrava", Zagreb, Zagreb
  - University of Zagreb School of Dental Medicine, Zagreb

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colorado-Bonnin M, Valmaseda-Castellon E, Berini-Aytes L, Gay-Escoda C. Quality of life following lower third molar removal. Int J Oral Maxillofac Surg. 2006 Apr;35(4):343-7. doi: 10.1016/j.ijom.2005.08.008. Epub 2005 Nov 8. PMID 16280233
- [Background] Borazan H, Kececioglu A, Okesli S, Otelcioglu S. Oral magnesium lozenge reduces postoperative sore throat: a randomized, prospective, placebo-controlled study. Anesthesiology. 2012 Sep;117(3):512-8. doi: 10.1097/ALN.0b013e3182639d5f. PMID 22797283
- [Background] Wilimzig C, Latz R, Vierling W, Mutschler E, Trnovec T, Nyulassy S. Increase in magnesium plasma level after orally administered trimagnesium dicitrate. Eur J Clin Pharmacol. 1996;49(4):317-23. doi: 10.1007/BF00226334. PMID 8857079
- [Background] Nicar MJ, Pak CY. Oral magnesium load test for the assessment of intestinal magnesium absorption. Application in control subjects, absorptive hypercalciuria, primary hyperparathyroidism, and hypoparathyroidism. Miner Electrolyte Metab. 1982 Jul;8(1):44-51. PMID 6897741
- [Background] Koseoglu E, Talaslioglu A, Gonul AS, Kula M. The effects of magnesium prophylaxis in migraine without aura. Magnes Res. 2008 Jun;21(2):101-8. PMID 18705538
- [Background] Bagis S, Karabiber M, As I, Tamer L, Erdogan C, Atalay A. Is magnesium citrate treatment effective on pain, clinical parameters and functional status in patients with fibromyalgia? Rheumatol Int. 2013 Jan;33(1):167-72. doi: 10.1007/s00296-011-2334-8. Epub 2012 Jan 22. PMID 22271372
- [Background] Walker AF, Marakis G, Christie S, Byng M. Mg citrate found more bioavailable than other Mg preparations in a randomised, double-blind study. Magnes Res. 2003 Sep;16(3):183-91. PMID 14596323
- [Background] Baqain ZH, Karaky AA, Sawair F, Khraisat A, Duaibis R, Rajab LD. Frequency estimates and risk factors for postoperative morbidity after third molar removal: a prospective cohort study. J Oral Maxillofac Surg. 2008 Nov;66(11):2276-83. doi: 10.1016/j.joms.2008.06.047. PMID 18940492
- [Background] Vormann J. Magnesium: nutrition and metabolism. Mol Aspects Med. 2003 Feb-Jun;24(1-3):27-37. doi: 10.1016/s0098-2997(02)00089-4. PMID 12537987
- [Derived] Jerkovic D, Tadin A, Gavic L, Vladislavic NZ, Grgic N, Macan D. Effect of orally administered magnesium on postoperative pain level and trismus after surgical removal of the lower third molars: a randomized, double-blind, placebo-controlled trial. Clin Oral Investig. 2020 Dec;24(12):4649-4659. doi: 10.1007/s00784-020-03335-z. Epub 2020 May 20. PMID 32436160